CLINICAL TRIAL: NCT01513382
Title: Does Intraoperative Methylene Blue Guidance in Pilonidal Sinus Surgery Really Effective in Total Excision of the Nest ?
Brief Title: Effectiveness of Methylene Blue Guidance in Total Excision of Pilonidal Sinus.
Acronym: BAVUGC-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Suleyman Bozkurt, Medical Doctor, Bezmialem Vakif University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BAVUGC-2
Record Dates: First submitted 2012-01-17; First posted 2012-01-20 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Pilonidal Sinus
Keywords: Pilonidal sinus; Methylene blue; Histopathology; Surgery
MeSH Terms: conditions — Pilonidal Sinus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Methylene Blue (Experimental): The effect of methylene blue dye in detection and total excision of pilonidal sinus will be studied histopathologically.
  Interventions: Procedure: Pilonidal sinus excision

INTERVENTIONS:
Procedure: Pilonidal sinus excision — The dyed portion of the excised pilonidal sinus and non-dyed cavity excision specimen will be studied histopathologically to detect any remnant of pilonidal sinus.

SUMMARY:
Methylene bleu use in pilonidal sinus surgery is not an effective guidance as expected.

DETAILED DESCRIPTION:
To study the potential benefits of intraoperative methylene blue use in pilonidal sinus surgery in detecting the borders of the disease, the histopathologic correlation between the specimen dyed by methylene blue and also the cavity excision specimen not dyed by methylene blue was investigated. The branches that distinctly exceeded the planned dyed excision borders will tried to be detected histopathologically, if any.

ELIGIBILITY:
Inclusion Criteria:

* Pilonidal sinus disease of the intergluteal region
* Primary disease without history of drainage
* Ages between 18 and 65, both gender

Exclusion Criteria:

* Recurrent pilonidal sinus disease
* Acute infection with abscess formation and/or purulent copious drainage
* Denial to sign informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Histopathologic detection of any evidence of pilonidal sinus disease in the cavity excision material not dyed by methylene blue | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Suleyman Bozkurt, M.D., Principal Investigator — Bezmialem Vakif University, Faculty of Medicine, Department of Surgery; Erhan Aysan, Prof. Dr., Study Director — Bezmialem Vakif University, Faculty of Medicine, Department of Surgery
Locations (1):
- Bezmialem Vakif University, Faculty of Medicine, Department of Surgery, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Result] Doll D, Novotny A, Rothe R, Kristiansen JE, Wietelmann K, Boulesteix AL, Dusel W, Petersen S. Methylene Blue halves the long-term recurrence rate in acute pilonidal sinus disease. Int J Colorectal Dis. 2008 Feb;23(2):181-7. doi: 10.1007/s00384-007-0393-9. Epub 2007 Oct 25. PMID 17960395
- [Result] Soll C, Hahnloser D, Dindo D, Clavien PA, Hetzer F. A novel approach for treatment of sacrococcygeal pilonidal sinus: less is more. Int J Colorectal Dis. 2008 Feb;23(2):177-80. doi: 10.1007/s00384-007-0377-9. Epub 2007 Aug 17. PMID 17703314
- [Result] Mentes O, Oysul A, Harlak A, Zeybek N, Kozak O, Tufan T. Ultrasonography accurately evaluates the dimension and shape of the pilonidal sinus. Clinics (Sao Paulo). 2009;64(3):189-92. doi: 10.1590/s1807-59322009000300007. PMID 19330243